CLINICAL TRIAL: NCT03605030
Title: Reducing Radiation Exposure to Operators During Invasive Cardiac Procedures With a Novel Lead-Based Arm-Board
Brief Title: Reducing Radiation Exposure to Operators During Invasive Cardiac Procedures
Acronym: RADAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Collaborators: Western University, Canada (Other)
Responsible Party: Principal Investigator, Pallav Garg, Assistant Professor, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 108913
Record Dates: First submitted 2018-07-21; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Patients Undergoing Invasive Cardiac Procedures; Radiation Exposure
Keywords: Cardiac Catheterization; Percutaneous Coronary Intervention; Radiation; Lead Shielding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel Lead Based Armboard (Active Comparator)
  Interventions: Device: Novel Lead Based Armboard
- Standard Armboard (Placebo Comparator)
  Interventions: Device: Standard Armboard

INTERVENTIONS:
Device: Novel Lead Based Armboard — Novel Lead Based Armboard
  Arms: Novel Lead Based Armboard
Device: Standard Armboard — Standard Armboard (without lead)
  Arms: Standard Armboard

SUMMARY:
The primary objective of this study is to determine if a novel lead-based arm board is effective at reducing radiation dose to the operator during invasive cardiac procedures. Secondary objectives are to measure effect on radiation dose to patient and total fluoroscopy (x-ray) time.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Planned invasive cardiology procedure, cardiac catheterization with or without percutaneous coronary intervention (PCI), or PCI alone.

Exclusion Criteria:

* Inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Radiation dose (μSv) to the operator at the chest | At procedure completion
  Co-primary outcomes included radiation dose (μSv; mean ± SD) to the operator at the chest and forearm level.
Radiation dose (μSv) to the operator at the forearm level | At procedure completion
  Co-primary outcomes included radiation dose (μSv; mean ± SD) to the operator at the chest and forearm level.

SECONDARY OUTCOMES:
Air kerma | At procedure completion
Dose area product | At procedure completion
Radiation dose to the patient | At procedure completion

CONTACTS AND LOCATIONS:
Overall Officials: Pallav Garg, MBBS, MSc, Principal Investigator — London Health Sciences Centre, Western University, London, ON
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided